CLINICAL TRIAL: NCT04699578
Title: Impact of COVID-19 Infection on the Course of Pregnancy and Fetal-neonatal Outcomes
Brief Title: COVID-19 Infection and Fetal-neonatal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Maddalena Morlando, Assistant Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 8453
Record Dates: First submitted 2021-01-01; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Obstetric Complication; SARS-CoV Infection; Preterm Birth; Miscarriage; Placenta Diseases
Keywords: obstetric; Covid19; SARS-CoV Infection; placenta; preterm birth
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Premature Birth; Abortion, Spontaneous; Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab with rRT-PCR as per ministerial protocol and in any case repeated at any admission to the hospital ward
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Covid-19 positive — All pregnant women at any stage of pregnancy afferent to obstetrics services who tested positive in confirmation tests by nasopharyngeal swab for viral RNA detection through real-time reverse transcriptase - polymerase chain reaction (rRT-PCR) will be included.

SUMMARY:
COVID-19, the coronavirus responsible for the pandemic that began at the end of 2019 in China, spreads through respiratory droplets and direct contact. The most common symptoms of the disease include fever, cough, asthenia or myalgia, wheezing and headache, and the most serious complication is acute respiratory distress syndrome (ARDS). The new coronavirus has continued to spread to multiple countries and continents so much so that the epidemic was declared a Public Health Emergency of International Interest (PHEIC) by the World Health Organization (WHO) on January 30, 2020. In the first phase of emergency worldwide, characterized by high morbidity and mortality, scientific interest has been mainly directed to the study of the transmission mechanisms of the infection, diagnostic tools and therapies for ARDS, especially in elderly and co-morbid patients. Interest has rapidly spread to other categories of patients and in particular to pregnancy, on which the virus could impact in different ways, with consequences for both the mother and the fetus. A recent systematic review that included all published reports on Coronaviruses (COVID-19, SARS, and MERS) in pregnancy showed that preterm delivery is the most frequently reported adverse event in these women, and that COVID-19 is associated with an increased risk of preeclampsia and caesarean section. Nonetheless, the limited sample size, the main inclusion of cases reported for acute respiratory symptoms, the lack of information on previous pathologies potentially capable of complicating pregnancy, do not allow for the extrapolation of strong evidence on the course of infection in pregnancy. Therefore, the current status of the scientific literature does not allow for general and wide-ranging implications. THe investigators therefore believe it is particularly useful to investigate maternal and fetal outcomes in this new broader scenario, including all pregnancies associated with asymptomatic or symptomatic SARS-CoV-2 infection, found in any gestational period, in order to evaluate in a "real world scenario" "Actual rates of maternal-fetal and neonatal adverse events

DETAILED DESCRIPTION:
Coronaviruses are a large family of viruses known to cause illnesses ranging from the common cold to more serious illnesses such as Middle East Respiratory Syndrome (MERS) and Severe Acute Respiratory Syndrome (SARS). They are positive-stranded RNA viruses, with a corona-like appearance under the electron microscope, whose primary target cells are the epithelial cells of the respiratory and gastrointestinal tract. The 2019/20 COVID-19 respiratory disease pandemic, caused by a coronavirus, began in December 2019 in the city of Wuhan, the capital of the Chinese province of Hubei, which has subsequently spread to several countries around the world. In early January 2020, health authorities identified the virus responsible for the epidemic, designating it, initially as "Coronavirus 2019-nCoV" but later with the official name of "SARS-CoV-2". To date, seven Coronaviruses have been shown to be capable of infecting humans: Common Human Coronaviruses: HCoV-OC43 and HCoV-HKU1 (Betacoronavirus) and HCoV-229E and HCoV-NL63 (Alphacoronavirus); they can cause common colds but also severe lower respiratory tract infections; other human coronaviruses (Betacoronaviruses): SARS-CoV, MERS-CoV and 2019-nCoV (now referred to as SARS-CoV-2).

SARS-CoV-2 is therefore the seventh virus of the same family that involves humans, spreads through respiratory droplets and direct contact. The most common symptoms of the disease include fever, cough, asthenia or myalgia, wheezing and headache, and the most serious complication is acute respiratory distress syndrome (ARDS). The new coronavirus has continued to spread to multiple countries and continents so much so that the outbreak was declared a public health emergency of international concern (PHEIC) by the World Health Organization (WHO) on January 30, 2020.

In the first phase of world emergency, characterized by high morbidity and mortality, scientific interest has been mainly focused on the study of the transmission mechanisms of the infection, diagnostic tools and therapies for ARDS, especially in elderly patients and with co-morbidities. Interest has rapidly spread to other categories of patients and in particular to pregnancy, on which the virus could impact in different ways, with consequences for both the mother and the fetus.

During pregnancy, different changes in the immune system and adaptive changes affecting organs and systems are observed in relation to the gestational period, among which those affecting the respiratory system are highlighted, particularly evident in the third trimester including, upper airway mucosal edema induced by elevated levels of estrogen and progesterone, elevation of the diaphragm and consequent limited lung expansion, and high oxygen consumption, all conditions that increase the susceptibility of pregnant women to respiratory insults.

The maternal immune system during pregnancy undergoes specific adaptations aimed at establishing and maintaining a fetal allogeneic tolerance while preserving the ability to protect against external infectious agents. It goes from a pro-inflammatory state in the first trimester (important for implantation and placentation) to an anti-inflammatory state in the second trimester (necessary for fetal growth), and finally returns to a pro-inflammatory state again in the third trimester and during childbirth. In addition, innate immunity cells, that is, NK cells and monocytes respond more actively to viral insults, while the adaptive immune response is down-regulated (Hong Liu et al). As for CD4 + (Th) T cells, involved in the regulation of the inflammatory response through the production of cytokines, there is a shift in the maternal immune response from Th1 (with pro-inflammatory action) towards Th2 (with anti-inflammatory action ), a crucial modification for maintaining maternal-fetal tolerance (Wegmannetal et al.).

In the first phase of world emergency, characterized by high morbidity and mortality, scientific interest has been mainly focused on the study of the transmission mechanisms of the infection, diagnostic tools and therapies for ARDS, especially in elderly patients and with co-morbidities. Interest has rapidly spread to other categories of patients and in particular to pregnancy, on which the virus could impact in different ways, with consequences for both the mother and the fetus.

During pregnancy, different changes in the immune system and adaptive changes affecting organs and systems are observed in relation to the gestational period, among which those affecting the respiratory system are highlighted, particularly evident in the third trimester including, upper airway mucosal edema induced by elevated levels of estrogen and progesterone, elevation of the diaphragm and consequent limited lung expansion, and high oxygen consumption, all conditions that increase the susceptibility of pregnant women to respiratory insults.

It is widely demonstrated that maternal systemic infections, which cause instability in the delicate balance of the immune system, may be related to the onset of complications during pregnancy, such as increased risk of miscarriage, intrauterine growth retardation, death fetal intrauterine.

Based on these pathophysiological assumptions, it is conceivable that SARS-CoV-2 infection could clinically modify the course of pregnancy and lead to fetal-neonatal complications.

Recent studies in the literature have shown that severe forms of COVID-19 disease are associated with a cytokine storm, characterized by increased concentrations of IL-2, IL-7, IL-10, G-CSF (granulocyte-colony stimulating factor), interferon-γ-inducible protein, MCP (monocyte chemoattractant protein), MIP- α (macrophage inflammatory protein alpha) and TNF α (tumor necrosis factor α). It has been hypothesized that during pregnancy this cytokine cascade could induce an even more severe inflammatory state, particularly in the first and third trimester of pregnancy (Hong Liu et al).

Recently, Ashary et al. analyzed the possible presence of the virus at the level of the syncytiotrophoblast, noting that in 12% of patients with active COVID-19 infection, the virus was identifiable at the placental level. Furthermore, the target receptors of the virus for entry into the cell, ACE-2 and TMPRSS2, are significantly expressed and used by the virus also at the placental level, so SARS-CoV-2 could potentially, interacting with these targets, alter the syncytiotrophoblastic unit and, consequently, the placental function (Seethy et al.)

Although the current evidence does not support a vertical intrauterine transmission of coronaviruses (Chen et al), it is likely that it is the same maternal infection and the inflammatory state in the course of the disease that can negatively influence the maternal-fetal outcome.

Given the multiple characteristics common to SARS-CoV1, MERS and SARS-CoV2 infections, of particular relevance were the studies conducted by Wong et al on SARS-CoV-1 infection in the first trimester, in which four out of seven women ( 57%), who contracted SARS during the first trimester, then had a miscarriage, and that of Alfaraj et al on MERS infection, in which there was a single case of a woman with MERS in the first trimester, who never developed symptoms of the disease, and carried the pregnancy to term.

A recent systematic review that included all published reports on Coronaviruses (COVID-19, SARS, and MERS) in pregnancy showed that preterm delivery is the most frequently reported adverse event in these women, and that COVID-19 is associated with an increased risk of preeclampsia and caesarean section. Nevertheless, the limited sample size, the main inclusion of cases reported for acute respiratory symptoms, the absence of information on previous pathologies potentially capable of complicating pregnancy, do not allow to extrapolate strong evidence on the course of infection in pregnancy ( Di Mascio et al. 2020).

Recently, Ashary et al. analyzed the possible presence of the virus at the level of the syncytiotrophoblast, noting that in 12% of patients with active COVID-19 infection, the virus was identifiable at the placental level. Furthermore, the target receptors of the virus for entry into the cell, ACE-2 and TMPRSS2, are significantly expressed and used by the virus also at the placental level, so SARS-CoV-2 could potentially, interacting with these targets, alter the syncytiotrophoblastic unit and, consequently, the placental function (Seethy et al.)

Although the current evidence does not support a vertical intrauterine transmission of coronaviruses (Chen et al), it is likely that it is the same maternal infection and the inflammatory state in the course of the disease that can negatively influence the maternal-fetal outcome.

Given the multiple characteristics common to SARS-CoV1, MERS and SARS-CoV2 infections, of particular relevance were the studies conducted by Wong et al on SARS-CoV-1 infection in the first trimester, in which four out of seven women ( 57%), who contracted SARS during the first trimester, then had a miscarriage, and that of Alfaraj et al on MERS infection, in which there was a single case of a woman with MERS in the first trimester, who never developed symptoms of the disease, and carried the pregnancy to term.

At the moment there are no data in the literature on the impact of SARS-CoV-2 infection on early pregnancy as the data currently available in the literature concern women hospitalized in serious clinical conditions during the first wave of the March 2020 pandemic (Di Mascio et al.). Conversely, other studies report low seroconversion rates for the virus. Therefore, the current status of the scientific literature does not allow for general and wide-ranging implications (La Cour Freiesleben et al.).

Furthermore, easier access to tests for the identification of COVID-19 and the introduction by hospitals of universal screening for COVID-19 at patient admissions, make it easier to identify the proportion of positive asymptomatic women. which could be, like what happens in the general population, particularly relevant, as well as the proportion of women diagnosed and subsequently resolved of the infection during pregnancy.

The investigators therefore believe it is particularly useful to investigate maternal and fetal outcomes in this new broader scenario, including all pregnancies associated with asymptomatic or symptomatic SARS-CoV-2 infection, found in any gestational period, in order to evaluate in a "real world scenario" "Actual rates of maternal-fetal and neonatal adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age> 18 years
* Women with single or multiple pregnancy at any stage of gestation, with first ascertained positivity to the nasopharyngeal swab for SARS-CoV-2 during pregnancy, regardless of the presence of symptoms.

Exclusion Criteria:

* age under 18.
* Women with an altered state of consciousness, seriously ill, with mental handicaps;
* Women with serious systemic diseases that can negatively affect the pregnancy outcome.
* Women for whom the treating doctor contraindicates participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All pregnant women at any stage of pregnancy afferent to obstetrics services who tested positive in confirmation tests by nasopharyngeal swab for viral RNA detection through real-time reverse transcriptase - polymerase chain reaction (rRT-PCR) will be included.
  Upon confirmation, women will be placed in a specific pregnancy monitoring program that will be defined as "at risk for SARS-COVID2", regardless of participation in this study. For women recruited in the study, no additional instrumental or laboratory investigations are required to be performed in addition to those already provided for in the normal clinical management of COVID-positive patients.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Preterm birth rate | Less than 37 weeks gestation

SECONDARY OUTCOMES:
Gestational age at delivery | Time of delivery
Preterm birth rates | Less than 24, 28, 34 weeks gestation
Birth weight | Time of delivery
  Weight of the baby at the time of delivery
Composite adverse neonatal outcomes | Between birth and 28 days of age
  Number of neonates who will have at least one of the following:
  necrotizing enterocolitis (NEC), intraventricular hemorrhage (IVH) (grade 3 or higher), respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD), retinopathy (ROP), blood-culture proven sepsis and neonatal death
Maternal outcomes | Between birth and 28 days after the birth
  Number of mothers who will have at least one of the following:
  sepsis, histological chorioamnionitis, hysterectomy, intensive care unit admission.
Inflammatory markers: coagulation profile, C-reactive protein, glycaemia, ferritinemia | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Colacurci, Professor, Study Director — University of Campania Luigi Vanvitelli; Fabiana Savoia, Study Chair — University of Campania Luigi Vanvitelli; Alessandra Familiari, Principal Investigator — Università Cattolica del Sacro Cuore - Dipartimento scienze della salute della donna e del bambino; Antonio Lanzone, Professor, Study Director — Università Cattolica del Sacro Cuore - Dipartimento scienze della salute della donna e del bambino; Antonio Schiattarella, MD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy